CLINICAL TRIAL: NCT04063267
Title: Electronic Cigarettes as a Harm Reduction Strategy in Individuals With Substance Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-00840
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Cigarette Smoking; Addiction; E Cig Use
MeSH Terms: conditions — Cigarette Smoking; Behavior, Addictive; Vaping | interventions — Electronic Nicotine Delivery Systems; Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E cigarettes (Experimental)
  Interventions: Other: E cigarettes
- Nicotine Replacement Therapy (Active Comparator)
  Interventions: Other: Nicotine Replacement Therapy

INTERVENTIONS:
Other: E cigarettes — Participants will be encouraged to substitute e-cigarettes for combustible cigarettes in order to reduce nicotine withdrawal symptoms
  Arms: E cigarettes
Other: Nicotine Replacement Therapy — Nicotine patches and gum to last them the first week based on their baseline recorded smoking. Participants will be advised to use both a 21 mg nicotine patch and 4 mg nicotine for cravings.
  Arms: Nicotine Replacement Therapy

SUMMARY:
Patients in addiction treatment have exceptionally higher rate of cigarette smoking and very low quit rates compared to the general population. The purpose of this study is to examine the feasibility of using e-cigarettes as a method for harm reduction and the effects of providing e-cigarettes (or placebo e-cigarettes) on smoking outcomes among patients in addiction treatment.

DETAILED DESCRIPTION:
Electronic nicotine delivery devices often referred to as e-cigarettes, are battery-powered devices that deliver vaporized nicotine when inhaled. Corresponding with the growth in media attention, marketing and promotion, awareness and use of e-cigarettes has increased dramatically. A large proportion of those using e-cigarettes use them to reduce the number of cigarettes they are smoking or to help them quit. Use of an e-cigarette by smokers unwilling or unable to stop smoking completely might be a good approach to reducing cigarette consumption as the e-cigarette imitates some behavioral aspects of cigarette smoking and contains nicotine. Moreover, the few existing studies on the effect of e-cigarettes on tobacco withdrawal and craving suggest promising potential to assist smokers in coping with smoking urges and decreasing cigarette use.

ELIGIBILITY:
Inclusion Criteria:

* smokes at least 10 cigarettes per day
* meet DSM-V AUD and/or OUD within the past year, interested in reducing CPDs
* able to provide consent
* use a cell phone, are willing/able to receive and respond to daily text messages regarding their cigarette use and e-cigarette use on their cell phone
* provide one additional contact, and are willing to use an e-cigarette for 3 weeks.

Exclusion Criteria:

* pregnant and/or breast feeding (self-reported)
* currently using smoking cessation medications (including other forms of NRT, buproprion, or varenicline)
* enrolled in a smoking cessation program or another cessation tria
* have used an e-cigarette in the past 14 days
* have used any other tobacco products (pipe, cigar, cigarillos, snuff, chewing tobacco, rolling tobacco, or hookah/shisha) in the past 30 days
* report having a history of asthma, other airways diseases, or heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who achieve 50% reduction in CPD at 3 weeks. | 3 Weeks
  proportion of participants who achieve 50% reduction in CPD at 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sherman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Scott.Sherman@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.